CLINICAL TRIAL: NCT01770015
Title: Study of the Impact of Bronchial Colonization With Fungi in the Occurrence of Late Ventilator Acquired Pneumonia
Brief Title: Bronchial Colonization With Fungi and Late Respiratory Acquired Pneumonia
Acronym: CBF et PAVMt
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Principal Investigator, AdministrateurDRC, Pr JF TIMSIT, University Hospital, Grenoble
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2011-A00767-34
Record Dates: First submitted 2012-06-21; First posted 2013-01-17 (Estimated); Last update posted 2022-11-04 (Actual); Status verified 2022-11

CONDITIONS: Ventilator Acquired Pneumonia
Keywords: patient ventilated for at least five days
MeSH Terms: conditions — Pneumonia, Ventilator-Associated | interventions — Cordocentesis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- ventilated patient (Experimental): all patients underwent the same diagnostic test . cutaneous, rectal, nose and mouth swabs to identify potential fungi colonization.
  HLA DR antigen, cytokines (IL 6 and 10), B-glucan. fungi and bacteria endotracheal aspiration
  Interventions: Procedure: biological sampling; Procedure: sampling blood; Procedure: endotracheal aspiration

INTERVENTIONS:
Procedure: biological sampling — cutaneous, rectal, nose and mouth swabs to identify potential fungi colonization
Procedure: sampling blood — HLA DR antigen, cytokines (IL 6 and 10), B-glucan
Procedure: endotracheal aspiration — fungi and bacteria endotracheal aspiration

SUMMARY:
Ventilator acquired pneumonia (VAP) are severe nosocomial infections. On the other side, bronchial fungi colonization is commonly observed in ICU; therefore, the investigators propose to study the role of bronchial fungi colonization on the occurrence of VAP taking into account the immune status of the patient and the antibiotic and antifungal treatments he has received.

ELIGIBILITY:
Inclusion Criteria:

* patient ventilated for at least 5 days

Exclusion Criteria:

* invasive infection Candida sp defined by : candidemia, isolation of Candida from a normally sterile site, candida pneumoniae.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 213 (Actual)
Dates: Start 2011-11; Primary Completion 2016-03 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Onset of a late ventilator acquired pneumonia (VAP) | Participants will be followed for the duration of mechanical ventilation, an expected time frame that can go from 5 days to up to 8 weeks

SECONDARY OUTCOMES:
Onset of a pseudomonas aeruginosa associated VAP | Participants will be followed for the duration of mechanical ventilation, an expected time frame that can go from 5 days to up to 8 weeks
Onset of late ventilator associated pneumonia associated to staphylococcus aureus | Participants will be followed for the duration of mechanical ventilation, an expected time frame that can go from 5 days to up to 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: TIMSIT Jean-François, PU/PH, Principal Investigator — University Hospital, Grenoble
Locations (2):
- France (2):
  - Hospital University Clermont Ferrand Gabriel Montpied, Clermont-Ferrand
  - University Hospital of Grenoble, Grenoble

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Timsit JF, Schwebel C, Styfalova L, Cornet M, Poirier P, Forrestier C, Ruckly S, Jacob MC, Souweine B. Impact of bronchial colonization with Candida spp. on the risk of bacterial ventilator-associated pneumonia in the ICU: the FUNGIBACT prospective cohort study. Intensive Care Med. 2019 Jun;45(6):834-843. doi: 10.1007/s00134-019-05622-0. Epub 2019 Apr 24. PMID 31020361